CLINICAL TRIAL: NCT03818295
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Praliciguat ([14C]-IW-1973) Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Trial to Study the Absorption, Metabolism, and Excretion of [14C]-Praliciguat in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRL-105
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Male Volunteers (Experimental): Single oral dose of [14C]-praliciguat
  Interventions: Drug: [14C]-praliciguat

INTERVENTIONS:
Drug: [14C]-praliciguat — 10 mg praliciguat containing approximately 500 μCi of [14C]-praliciguat
  Other Names: [14C]-IW-1973

SUMMARY:
The primary objective is to characterize the pharmacokinetics (PK) of praliciguat and total radioactivity and to assess the elimination of total radioactivity from a single oral dose of [14C]-praliciguat.

ELIGIBILITY:
Inclusion Criteria:

* Males of any race, between 18 and 55 years of age, inclusive
* Body mass index between 18 and 32 kg/m2, inclusive
* Subject is in good health and has no clinically significant findings on physical examination
* Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and for at least 90 days after the final dose of study drug

Exclusion Criteria:

* Any active or unstable clinically significant medical condition
* Use of any prescribed or non-prescribed medication

Additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Amount of total radioactivity excreted in urine (Aeu) and feces (Aef) | up to Day 15
Cumulative Aeu and cumulative Aef | up to Day 15
Percentage of total radioactivity excreted in urine (feu) and feces (fef) | up to Day 15
Cumulative feu and cumulative fef | up to Day 15
Percentage of total radioactivity in total excreta (feces + urine) | up to Day 15
Area under the concentration-time curve (AUC) from time zero to infinity (AUC0-inf) of praliciguat in plasma | up to Day 15
AUC0-inf of total radioactivity in plasma and whole blood | up to Day 15
AUC from time zero to the last quantifiable concentration (AUC0-last) of praliciguat in plasma | up to Day 15
AUC0-last of total radioactivity in plasma and whole blood | up to Day 15
Maximum observed concentration (Cmax) of praliciguat in plasma | up to Day 15
Cmax of total radioactivity in plasma and whole blood | up to Day 15
Time of Cmax (Tmax) of praliciguat in plasma | up to Day 15
Tmax of total radioactivity in plasma and whole blood | up to Day 15
Apparent terminal elimination half-life (t1/2) of praliciguat in plasma | up to Day 15
t1/2 total radioactivity in plasma and whole blood | up to Day 15
Apparent total clearance of praliciguat (CL/F) | up to Day 15
Apparent volume of distribution of praliciguat (Vz/F) | up to Day 15
AUC0-inf of plasma praliciguat concentration relative to AUC0-inf of plasma total radioactivity (AUC0-inf Ratio of Plasma Praliciguat/Plasma Total Radioactivity) | up to Day 15
AUC0-inf of whole blood total radioactivity to AUC0-inf of plasma total radioactivity (AUC0-inf Ratio of Blood Total Radioactivity/Plasma Total Radioactivity) | up to Day 15

SECONDARY OUTCOMES:
Levels of metabolite radioactivity excreted in urine and feces | up to Day 15
AUC0-inf of metabolite radioactivity levels in plasma | up to Day 15
AUC0-inf of plasma metabolite radioactivity levels relative to AUC0-inf of plasma total radioactivity (Plasma AUC0-inf Ratio of Metabolite Radioactivity/Total Radioactivity) | up to Day 15
Chromatographic retention time of metabolites | up to Day 15
Molecular ion mass of metabolites | up to Day 15
Characteristic mass spectrometry fragmentation ions of metabolites | up to Day 15
Chemical structures (graphical representations showing atom connectivity) proposed for plasma, urine, and feces metabolites | up to Day 15
Number(s) of participants with ≥1 treatment-emergent serious adverse event (SAE) | up to Day 15
Number(s) of participants with ≥1 adverse event (AE) leading to study drug discontinuation | up to Day 15
Number(s) of participants with ≥1 Grade ≥3 AE (per CTCAE v. 5.0) | up to Day 15
Number(s) of participants with ≥1 clinically significant abnormal physical examination finding | up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: John Hanrahan, MD, Study Director — Ironwood Pharmaceuticals, Inc.
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No